CLINICAL TRIAL: NCT05319015
Title: A Phase II Study of the Safety and Efficacy of Neoadjuvant Lenvatinib and Pembrolizumab in Patients With Renal Cell Carcinoma and IVC Tumor Thrombus
Brief Title: Neoadjuvant Lenvatinib and Pembrolizumab for IVC Tumor Thrombus
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Vitaly Margulis, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2021-1240
Record Dates: First submitted 2022-03-23; First posted 2022-04-08 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; IVC tumor thrombus; Neoadjuvant therapy; Immunotherapy; Nephrectomy
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Patients receive neoadjuvant lenvatinib (20 mg PO daily) for 12 weeks and pembrolizumab (200 mg IV every 3 weeks for four doses) prior to surgical resection of locally advanced RCC with IVC tumor thrombus. Following surgery, patients will receive adjuvant pembrolizumab (200 mg IV every 3 weeks for up to thirteen doses).
  Interventions: Drug: Neoadjuvant Lenvatinib; Drug: Neoadjuvant Pembrolizumab; Procedure: Radical nephrectomy, IVC thrombectomy, retroperitoneal lymph node dissection; Drug: Adjuvant Pembrolizumab

INTERVENTIONS:
Drug: Neoadjuvant Lenvatinib — 20 mg PO daily for 12 weeks prior to surgery
Drug: Neoadjuvant Pembrolizumab — 200 mg IV every 3 weeks for 4 doses prior to surgery
Procedure: Radical nephrectomy, IVC thrombectomy, retroperitoneal lymph node dissection — Resection of locally advanced RCC with IVC tumor thrombus
Drug: Adjuvant Pembrolizumab — 200 mg IV every 3 weeks for up to 13 doses after surgery

SUMMARY:
This study will be evaluating safety and efficacy of the combination of lenvatinib and pembolizumab neoaadjuvant therapy prior to surgical resection of locally advanced renal cell carcinoma with IVC tumor thrombus.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent
2. Have histologically confirmed cT3-4,N0-1,M0-1 (clinical stage III-IV) diagnosis of renal cell carcinoma (any subtype) with level II-IV inferior vena cava tumor thrombus as per the Mayo classification of macroscopic venous invasion in renal cell carcinoma:

   1. Level 1 tumor thrombus is either at the entry of renal vein or within the IVC < 2 cm from the confluence of renal vein and IVC
   2. Level II tumor thrombus extends within the IVC > 2 cm above the confluence of renal vein and IVC, but still remains below the hepatic veins.
   3. Level III tumor Thrombus involves the intrahepatic IVC.
   4. Level IV tumor thrombus extends above diaphragm or into the right atrium.
3. The primary tumor and thrombus may be assessed to be resectable or unresectable at the time of enrollment.
4. Male participants:

   A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the 120 day neoadjuvant treatment period and for at least 90 days after the last dose of study treatment and refrain from donating sperm during this period.

   Female participants:

   A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:
   1. Not a woman of childbearing potential (WOCBP) OR
   2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 30 days after the last dose of study treatment.
5. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
6. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
7. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 14 days prior to the first dose of study intervention.
8. Criteria for known Hepatitis B and C positive subjects

   Hepatitis B and C screening tests are not required unless:
   * Known history of HBV or HCV infection
   * As mandated by local health authority

   Hepatitis B positive subjects:

   Participants who are HBsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization. Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention.

   Hepatitis C positive subjects:

   Participants with history of HCV infection are eligible if HCV viral load is undetectable at screening.
9. Participants must have completed curative anti-viral therapy at least 4 weeks prior to randomization
10. HIV-positive participants may be enrolled.
11. HIV-infected participants must have well-controlled HIV on ART, defined as:

1. Participants on ART must have a CD4+ T-cell count ≥350 cells/mm3 at the time of screening 2. Participants on ART must have achieved and maintained virologic suppression defined as confirmed HIV RNA level below 50 or the LLOQ (below the limit of detection) using the locally available assay at the time of screening and for at least 12 weeks before screening 3. It is advised that participants must not have had any AIDS-defining opportunistic infections within the past 12 months.

4. Participants on ART must have been on a stable regimen, without changes in drugs or dose modification, for at least 4 weeks before study entry (Day 1) and agree to continue ART throughout the study 5. The combination ART regimen must not contain any antiretroviral medications that interact with CYP3A4 inhibitors/inducers/substrates (https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers)

12. Have adequate organ function as defined in the following table (Table 4). Specimens must be collected within 14 days prior to the start of study intervention.

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
3. Has received prior systemic anti-cancer therapy including investigational agents prior to allocation.
4. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
5. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed. COVID-19 vaccines are permitted provided they are not live attenuated vaccines.
6. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention with the exception of participating in the exploratory imaging trial utilizing 89Zr-DFO-Atezolizumab ImmunoPET/CT (STU-2019-0714).
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. Has a known additional malignancy that is progressing or has required active treatment within the past year. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (eg, breast carcinoma, cervical cancer, bladder in situ) that have undergone potentially curative therapy are not excluded.
9. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
10. Has more than three different sites of metastatic renal cell carcinoma.
11. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and lenvatinib and/or any of its excipients.
12. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
13. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
14. Has an active infection requiring systemic therapy.
15. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
16. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
17. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
18. Has had an allogenic tissue/solid organ transplant.
19. Has prolongation of QTcF interval to >480 ms.
20. Has a left ventricular ejection fraction (LVEF) below the institutional (or local laboratory) normal range, as determined by multigated acquisition (MUGA) or echocardiogram (ECHO).

    1. Patients with an ejection fraction (LVEF) of 50 or greater are eligible to enroll on the study
    2. Patients with an ejection fraction (LVEF) of 40 to 49 are eligible to enroll on the study if they they DO NOT have signs of New York Heart Association Class III or IV congestive heart failure:

    i. NYHA Class III signs of congestive heart failure include marked limitation of physical activity - ordinary activity or movements cause significant fatigue, heart palpitations, or shortness of breath ii. NYHA Class IV signs of congestive heart failure include being unable to carry out physical activity without discomfort, having symptoms of heart failure at rest, if physical activity or movement is undertaken, discomfort increase c. Patients with an ejection fraction (LVEF) of 39 or less are not eligible to enroll on the study.
21. Has clinically significant cardiovascular disease within 12 months from first dose of study intervention, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability. Note: Medically controlled arrhythmia would be permitted.
22. If urinalysis reveals proteinuria of 2+ or 500mg/dL greater based on the scale below, the patient will need to undergo a 24 hour urine collection, if the patient has 2000mg/24 hour or great of protein in the 24 hour the urine collection they are NOT ELIGIBLE for the study. If urinalysis protein is negative, trace, 1+, or urinalysis protein is reported in the range 0-499mg/dL protein, the patient IS ELIGIBLE to enroll on the study and does not need to complete a 24 hour urine collection:

    1. 1+ = 200 - 500 mg/24 hours
    2. 2+ = 500 - 1500 mg/24 hours
    3. 3+ = over 2500 mg/24 hours
    4. 4+ = over 3000 mg/24 hours.
23. Uncontrolled blood pressure defined as consistently elevated blood pressure with a Systolic BP>140 mmHg or diastolic BP >90 mmHg in spite of an optimized regimen of antihypertensive medication are not able to enroll on the study. However, patients with borderline, isolated, or occasional elevation of blood pressure readings are eligible to enroll on the trial. If the treating physician believes the blood pressure elevation is transient the patient may enroll and blood pressure will be monitored during the study. Patients with persistent hypertension may be initiated on antihypertensive medication by the treating physician if deemed necessary and may enroll on the study. The treating physician may also adjust antihypertensive medication in the attempt to achieve a normal blood pressure while the patient is in screening and on study. It is at the discretion of the enrolling physician to continue adjusting the hypertension medication while the patient is enrolled and treated on the study to maintain adequate blood pressure readings.
24. HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease.
25. Patients with active Hepatitis B infection (defined as HBsAg positive and/or detectable HBV DNA).
26. Patients with active Hepatitis C infection (defined as anti-HCV Ab positive and detectable HCV RNA).
27. Hepatitis B and C screening tests are not required unless there is a known history of HBV and HCV infection or as mandated by local health authority.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-06 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate | 12 weeks
  Evaluation of changes in size of primary tumor and size and level of IVC tumor thrombus on imaging due to neoadjuvant therapy prior to surgery.
Local and Metastatic Progression Rate | 12 weeks
  Evaluation of local or metastatic progression on imaging prior to surgery following neoadjuvant therapy.
90 Day Post-Operative Complications | 13 weeks
  Assessment of 90 day post-operative safety and morbidity of neoadjuvant therapy by evaluating the incidence of 90 day post-operative grade 3-5 adverse events.

SECONDARY OUTCOMES:
Estimated blood loss | 1 week
  Estimated blood loss in mL during surgery
Operative time | 1 week
  Operative time in minutes of surgery, length of stay, and intra-operative and post-operative complications
Length of stay | 1 week
  Length of stay of hospital stay for surgery in days, and intra-operative and post-operative complications
Intra-operative complications | 1 week
  Complications that occur during surgery
Post-operative complications | 12 weeks
  Complications that occur in the post-operative period
Survival Outcomes | 3 years
  Evaluation of post-operative survival outcomes including recurrence-free survival and overall survival.

OTHER OUTCOMES:
Exploratory Outcomes | 24 weeks
  Identify metabolic signatures in plasma that are noninvasive predictors of therapy response and identify metabolic alterations following neoadjuvant therapy in patients who do and do not respond.

CONTACTS AND LOCATIONS:
Overall Officials: Vitaly Margulis, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No